CLINICAL TRIAL: NCT02465918
Title: The Relationship Between Cyclizing Stimulation and Effective Stimulation During Motor Cortex Stimulation
Brief Title: Cyclization of Motor Cortex Stimulation
Status: Completed | Phase: Not Applicable | Type: Interventional
Sponsor: University of British Columbia (Other)
Responsible Party: Principal Investigator, Christopher Honey, Associate Professor/Neurosurgeon, University of British Columbia
Allocation: Randomized | Model: Crossover | Masking: Single | Purpose: Treatment
Other Study IDs: H15-01420
Record Dates: First submitted 2015-06-04; First posted 2015-06-09 (Estimated); Last update posted 2020-10-30 (Actual); Status verified 2020-10

CONDITIONS: Neuropathic Pain
MeSH Terms: conditions — Neuralgia

STUDY DESIGN:
Who Masked: Participant
Oversight: Data Monitoring Committee: No

ARMS (4):
- Original Setting- MCS 30 min off/0 min off (Active Comparator): Patients at baseline with their original MCS settings: on 30 minutes, off 0 minutes in any single half-hour.
  Interventions: Device: motor cortex stimulation (Change of Stimulation Timing)
- MCS 25 min on/5 min off (Experimental): Patient MCS settings programmed to: on 25 minutes, off 5 minutes in any single half-hour.
  Interventions: Device: motor cortex stimulation (Change of Stimulation Timing)
- MCS 20 min on/10 min off (Experimental): Patient MCS settings programmed to: on 20 minutes, off 10 minutes in any single half-hour.
  Interventions: Device: motor cortex stimulation (Change of Stimulation Timing)
- MCS 15 min on/15 min off (Experimental): Patient MCS settings programmed to: on 15 minutes, off 15 minutes in any single hour.
  Interventions: Device: motor cortex stimulation (Change of Stimulation Timing)

INTERVENTIONS:
Device: motor cortex stimulation (Change of Stimulation Timing)

SUMMARY:
Motor cortex stimulation (MCS) is a form of brain stimulation for patients with neuropathic pain not responsive to medication. An electrode is placed on the surface of the brain and connected to a programmable battery in the chest.

The strength of stimulation can be individually adjusted by changing the voltage of stimulation. A too high voltage will produce side effects (e.g. seizures) while a too low voltage will not provide pain control.

The aim of this study is to analyze the optimal stimulation timing parameters in patients already implanted with MCS and have received good pain relief. The investigators wish to cyclize on/off MCS in order to save the battery life of the stimulator and also decrease stimulus habituation. The investigators hope to determine these timing parameters while maintaining optimal pain relief.

ELIGIBILITY:
Inclusion Criteria:

* Adult patient more than 18 years of age
* Chronic neuropathic pain effectively treated with motor cortex stimulation
* Stable medication during the trial
* Willing and able to comply with the study protocol and to return per the follow-up visit schedule and able to provide informed consent.

Exclusion Criteria:

* Evidence of an active disruptive psychiatric disorder or other known condition significant enough to impact the perception of pain, compliance to intervention and/or ability to evaluate treatment outcome as determined by the investigator
* Technical malfunction of the MCS device
* History of seizures
* Unable to provide informed consent

Min Age: 18 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 6 (Actual)
Dates: Start 2015-07; Primary Completion 2016-07 (Actual); Study Completion 2016-07 (Actual)

PRIMARY OUTCOMES:
Change in Pain measured on the Visual Analogue Scale (VAS) with different stimulation settings | At the End of each trial period, typically 14 days after change in stimulation settings

SECONDARY OUTCOMES:
Quality of Life assessment with the SF-36 questionnaire | At the end of each trial period, typically at 14 days after change in stimulation settings

OTHER OUTCOMES:
Pain assessment with the McGill pain questionnaire to record impact of pain | At the end of each trial period, typically 14 days after change in stimulation setting

CONTACTS AND LOCATIONS:
Locations (1):
- The Vancouver General Hospital, Vancouver, British Columbia, Canada

REFERENCES:
- [Result] Tsubokawa T, Katayama Y, Yamamoto T, Hirayama T, Koyama S. Treatment of thalamic pain by chronic motor cortex stimulation. Pacing Clin Electrophysiol. 1991 Jan;14(1):131-4. doi: 10.1111/j.1540-8159.1991.tb04058.x. PMID 1705329
- [Result] Tsubokawa T, Katayama Y, Yamamoto T, Hirayama T, Koyama S. Chronic motor cortex stimulation for the treatment of central pain. Acta Neurochir Suppl (Wien). 1991;52:137-9. doi: 10.1007/978-3-7091-9160-6_37. PMID 1792954
- [Result] Peyron R, Garcia-Larrea L, Deiber MP, Cinotti L, Convers P, Sindou M, Mauguiere F, Laurent B. Electrical stimulation of precentral cortical area in the treatment of central pain: electrophysiological and PET study. Pain. 1995 Sep;62(3):275-286. doi: 10.1016/0304-3959(94)00211-V. PMID 8657427
- [Result] Lima MC, Fregni F. Motor cortex stimulation for chronic pain: systematic review and meta-analysis of the literature. Neurology. 2008 Jun 10;70(24):2329-37. doi: 10.1212/01.wnl.0000314649.38527.93. PMID 18541887